CLINICAL TRIAL: NCT02613637
Title: Registry Study on Biological Disease Profile and Clinical Outcome in Patients With Newly Diagnosed or Existent Lung Cancer The LuCa Biology and Outcome (BiO)-Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Lars Bullinger, Prof. Dr., University of Ulm
Other Study IDs: LuCa BiO
Record Dates: First submitted 2015-06-22; First posted 2015-11-24 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; registry study; Biological Disease Profile
MeSH Terms: conditions — Lung Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — * Tumor tissue
  * 20-40 mL of peripheral blood in a heparinized (1:10) tube
  * 10 ml EDTA-anticoagulated blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry

SUMMARY:
Registry Study on Biological Disease Profile and Clinical Outcome in Patients with Newly Diagnosed or Existent Lung Cancer

The LuCa Biology and Outcome (BiO)-Project

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected diagnosis of lung cancer, or previously diagnosed lung cancer
* Age ≥ 18 years. There is no upper age limit.

Exclusion Criteria:

* Severe neurological or psychiatric disorder interfering with ability to give an informed consent
* No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician about study participation
* No consent for biobanking of patient's biological specimens and performance of analyses on stored material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed or existent lung cancer of all LuCa BiO centers in Germany are intended to be registered with in the LuCa BiO Registry.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-05; Primary Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | maximally 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bullinger, MD, Principal Investigator — University Hospital of Ulm
Locations (3):
- Germany (3):
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Pneumologie, Internistische Intensivmedizin, Beatmungsmedizin und Allgemeine Innere Medizin, Krankenhaus vom Roten Kreuz Bad Cannstatt GmbH, Stuttgart
  - Universitätsklinikum Ulm, Ulm